CLINICAL TRIAL: NCT04734691
Title: Second Line Oxaliplatin Based Chemotherapy Alone Versus Oxaliplatin Based PIPAC and Chemotherapy in Colorectal Peritoneal Carcinomatosis : A Phase II Randomize Mutli-centric Study : OPAC Study
Brief Title: Second Line Oxaliplatin Based Chemotherapy Alone Versus Oxaliplatin Based PIPAC and Chemotherapy in Colorectal Peritoneal Carcinomatosis : A Phase II Randomize Mutli-centric Study
Acronym: OPAC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sleiman Marwan-Julien (Other)
Responsible Party: Sponsor-Investigator, Sleiman Marwan-Julien, Doctor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPAC study
Record Dates: First submitted 2021-01-27; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Peritoneal Carcinomatosis
MeSH Terms: conditions — Peritoneal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental)
  Interventions: Procedure: PIPAC
- Control Arm (Active Comparator)
  Interventions: Procedure: PIPAC

INTERVENTIONS:
Procedure: PIPAC — PIPAC is a laparoscopic procedure for intraperitoneal administration of chemotherapy

SUMMARY:
Colorectal cancer is the third most common cancer in men and second in women. It represent 345'346 new cases per year in Europe and 134'349 in the United States of America. The peritoneal cavity is the second most frequent site, after liver, for colorectal cancer relapse.Peritoneal carcinomatosis (PC) is found in approximately 5 % of patients diagnosed with colorectal cancer and 24% of patients with synchronous metastasis at the time of diagnosis. Eight percent of colorectal cancer patient will develop PC during the course of their disease .

Currently systemic chemotherapy is the standard of care for the treatment of unresectable peritoneal carcinomatosis from colorectal cancer with a median survival rate of 16.3 months Peritoneal carcinomatosis has a poor response to systemic chemotherapy due to a weak penetration of agents into the peritoneum.

A new approach of intraperitoneal carcinomatosis is now developed: Pressurized intraperitoneal aerosol chemotherapy (PIPAC) is used to deliver intraperitoneal chemotherapy. It enhances the effect of chemotherapy because of the physical properties of aerosol and pressure.

PIPAC is a safe with a 23% morbidity and tolerated technic that is now well described.

We want to conduct a study to prove or infirm the superiority of PIPAC associated with systemic chemotherapy compare to systemic chemotherapy alone in peritoneal carcinomatosis from colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 < age ≤ 75 years old with Performance status (WHO) ≤ 2 Histologically evidenced synchronous or metachronous PM of a colorectal cancer with a PCI ≥ 15 (No complete resectable PC) Histologically evidenced synchronous or metachronous PM of a colorectal cancer with a PCI < 15 + liver or pulmonary unresectable metastases PCI < 15 but with progression at the restaging after the first line of chemotherapy Unresectable peritoneal relapse secondary to cytoreduction surgery

Exclusion Criteria:

* Patients with clinically significant ascites (> 3000 cc)
* Pleural effusion requiring evacuation for respiratory failure
* Small bowel occlusion with no possible food intake
* Presence of comorbidities, notably serious chronic diseases or organ failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 8 months
  any clinical sign and/or morphological sign of peritoneal recurrence or death

SECONDARY OUTCOMES:
Quality of life C30 | 8 months

IPD SHARING:
Plan to Share IPD: Undecided